CLINICAL TRIAL: NCT01921985
Title: Terlipressin Administration in Patients Undergoing Major Liver Resection: a Prospective Randomized Blinded Trial
Brief Title: Terlipressin Administration in Patients Undergoing Major Liver Resection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis revealed that no statistical difference will be identified after inclusion of the patient cohort as foreseen in the sample size calculation
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 190/11
Record Dates: First submitted 2013-08-09; First posted 2013-08-14 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Liver Resection; Liver Failure
MeSH Terms: conditions — Liver Failure | interventions — Terlipressin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Terlipressin (Active Comparator): Terlipressin given as intravenous injections of 1mg iv in 100ml of NaCl every 6 hours (total duration of drug administration 120 hours, cumulative dose is 20mg).
  Interventions: Drug: Terlipressin
- NaCl (Placebo Comparator): Placebo (Saline 100 ml) administered every 6 hours (total duration of drug administration 120 hours).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Terlipressin — Terlipressin given as intravenous injections of 1mg iv in 100ml of NaCl every 6 hours (total duration of drug administration 120 hours, cumulative dose is 20mg).
  Arms: Terlipressin
Drug: Placebo — Placebo (Saline 100 ml) administered every 6 hours (total duration of drug administration 120 hours).
  Arms: NaCl

SUMMARY:
This study investigates if the administration of terlipressin reduces complications after major liver surgery.

DETAILED DESCRIPTION:
Background

Surgery offers the only potential cure in many patients with primary or metastatic liver cancer. Extending the limits and improving safety of liver resection would allow more patients to benefit from surgery and to increase their survival. The prerequisite for successful and safe liver surgery is the optimal regeneration of the remaining hepatic tissue in order to fulfill the metabolic demands of the patient. Liver regeneration depends on a correct portal pressure and portal blood flow. In the preliminary results the investigators show an elevation of portal pressure post partial hepatectomy in mice. Pharmacologic reduction of such elevated portal pressure using terlipressin, a vasopressin agonist, was associated with improved liver regeneration.

Objective

Surgery offers the only potential cure in many patients with primary or metastatic liver cancer. Extending the limits and improving safety of liver resection would allow more patients to benefit from surgery and to increase their survival. Liver regeneration depends on a correct portal pressure and portal blood flow. Pharmacologic reduction of elevated portal pressure using terlipressin, a vasopressin agonist, is potentially associated with improved liver regeneration. Aim: To perform a prospective randomized trial comparing terlipressin versus placebo in patients undergoing major hepatic resection.

Methods

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing resection of 3 or more liver segments
* Minimum age of 18
* Any gender
* Written informed consent

Exclusion Criteria

* Preoperative renal failure (GFR < 50ml/min)
* Severe liver dysfunction (Child-Turcotte-Pugh grade C)
* Hyponatremia (<132mmol/l)
* Severe aortic regurgitation, severe mitral regurgitation, heart failure
* Symptomatic coronary heart disease
* Bradycardic arrhythmia (heart rate < 60/min)
* Peripheral artery occlusive disease (clinical stadium II-IV)
* Dilatative arteriopathy, history of subarachnoidal bleeding
* Decompensated arterial hypertension (Blood pressure >160/100mmHg despite intensive treatment)
* Present or suspected acute mesenteric ischemia
* Septic shock
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-11; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with incident of a composite end point | one month

SECONDARY OUTCOMES:
Number of patients with pleural effusion | one month
Number of patients with surgical site infection | one month
Number of patients with sepsis | one month
Number of patients with pneumonia | one month
Number of patients with intraabdominal hematoma | one month
Number of patients with acute renal failure | one month
Number of patients with blood transfusion | one month

CONTACTS AND LOCATIONS:
Overall Officials: Guido Beldi, Professor Dr. med., Principal Investigator — University of Bern
Locations (1):
- Dep. of Visceral Surgery, University Hospital Berne, Bern, Switzerland

REFERENCES:
- [Derived] Kohler A, Perrodin S, De Gottardi A, Candinas D, Beldi G. Effectiveness of terlipressin for prevention of complications after major liver resection - A randomized placebo-controlled trial. HPB (Oxford). 2020 Jun;22(6):884-891. doi: 10.1016/j.hpb.2019.10.011. Epub 2019 Oct 31. PMID 31680011